CLINICAL TRIAL: NCT03508947
Title: A Multicenter, Double-blind, Placebo-controlled, Phase 1 Study of WVE-210201 Administered Intravenously to Patients With Duchenne Muscular Dystrophy
Brief Title: Safety and Tolerability of WVE-210201 in Patients With Duchenne Muscular Dystrophy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wave Life Sciences Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: WVE-DMDX51-001
Record Dates: First submitted 2018-04-16; First posted 2018-04-26 (Actual); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Duchenne Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- WVE-210201 (Dose A) or placebo (Experimental)
  Interventions: Drug: WVE-210201; Drug: Placebo
- WVE-210201 (Dose B) or placebo (Experimental)
  Interventions: Drug: WVE-210201; Drug: Placebo
- WVE-210201 (Dose C) or placebo (Experimental)
  Interventions: Drug: WVE-210201; Drug: Placebo
- WVE-210201 (Dose D) or placebo (Experimental)
  Interventions: Drug: WVE-210201; Drug: Placebo
- WVE-210201 (Dose E) or placebo (Experimental)
  Interventions: Drug: WVE-210201; Drug: Placebo

INTERVENTIONS:
Drug: WVE-210201 — WVE-210201 is a stereopure antisense oligonucleotide (ASO)
Drug: Placebo — Sodium Chloride

SUMMARY:
This is a Phase 1, double-blind, placebo-controlled, single ascending dose cohort study to evaluate the safety, tolerability, and plasma concentrations of WVE-210201 in ambulatory and non-ambulatory male pediatric patients with DMD amenable to exon 51 skipping intervention.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Duchenne muscular dystrophy (DMD) based on clinical phenotype with increased serum creatine kinase
* Documented mutation in the Dystrophin gene associated with DMD that is amenable to exon 51 skipping
* Ambulatory or non-ambulatory male patients aged ≥5 - ≤18 years
* Stable pulmonary and cardiac function as measured by:

  1. Reproducible percent predicted forced vital capacity (FVC) ≥50%
  2. Left ventricular ejection fraction (LVEF) >55% in patients <10 years of age and >45% in patients ≥10 years of age, as measured (and documented) by echocardiogram within one year prior to enrollment into the study.

Exclusion Criteria:

* Severe cardiomyopathy; cardiomyopathy that is managed by angiotensin-converting enzyme (ACE) inhibitors or beta blockers is acceptable provided the patient meets the LVEF inclusion criteria.
* Need for mechanical or non-invasive ventilation OR anticipated need for mechanical or non-invasive ventilation within the next year, in the opinion of the Investigator.
* Changes in nutritional or herbal supplements or concomitant medications within 1 month prior to Screening visit or plans to modify dose or regimen during the study.
* Currently on anticoagulants or antithrombotics.
* Received treatment with eteplirsen or ataluren within the past 14 weeks.
* Received prior treatment with drisapersen.
* Received any investigational drug within the past 3 months or 5 half-lives, whichever is longer.

Ages: 5 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 36 (Actual)
Dates: Start 2018-01-24 (Actual); Primary Completion 2019-03-06 (Actual); Study Completion 2019-03-06 (Actual)

PRIMARY OUTCOMES:
Safety: Number of patients with adverse events (AEs) | Day 1 to Day 85 (end of study)
Safety: Severity of AEs | Day 1 to Day 85 (end of study)
Safety: Number of patients with serious AEs (SAEs) | Day 1 to Day 85 (end of study)
Safety and Tolerability: Number of patients who withdraw due to AEs | Day 1 to Day 85 (end of study)

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Maximum observed concentration (Cmax) | Day 1, Day 2, and Day 8
PK: Time of occurrence of Cmax (tmax) | Day 1, Day 2, and Day 8
PK: Area under the plasma concentration-time curve (AUC 0-t) | Day 1, Day 2, and Day 8

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Panzara, MD, MPH, Study Director — Wave Life Sciences Ltd.
Locations (13):
- Rare Disease Research, LLC., Atlanta, Georgia, United States
- Belgium (3):
  - UZ Gent, Ghent
  - Universitaire Ziekenhuizen Leuven, Leuven
  - CHR de la Citadelle, Liège
- London Health Sciences Centre - Hospital, London, Ontario, Canada
- Hôpital Armand Trousseau, Paris, France
- Italy (2):
  - U.O.C di Neurologia e Malattie Neuromuscolari Centro Clinico Nemo Sud, Messina
  - U.O. Immunologia Pediatrica, Milan
- Radbound University Nijmegen Medical Care, Nijmegen, Netherlands
- United Kingdom (4):
  - University Hospitals Bristol NHS Foundation Trust, Bristol
  - Alder Hey Children's Hospital, Liverpool
  - Evelina London Children's Hospital, London
  - UCL Institute of Child Health & Great Ormond Street Hospital for Children, London